CLINICAL TRIAL: NCT03610646
Title: A Multi Center, Randomized, Double-Masked, Active-Controlled, Comparative Clinical Study to Evaluate the Efficacy and Safety of MYL-1701P and Eylea® in Subjects With Diabetic Macular Edema (DME)
Brief Title: Comparative Study to Evaluate the Efficacy and Safety of MYL-1701P and Eylea® in Subjects With Diabetic Macular Edema (DME)
Acronym: DME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Collaborators: Momenta Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MYL-1701P-3001
Record Dates: First submitted 2018-07-09; First posted 2018-08-01 (Actual); Results first posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema,; BCVA,; ETDRS Letters.
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either MYL-1701P or Eylea groups in parallel for the duration of the study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Masked study drug kits will be supplied to sites as necessary during the study. The outside label of the box will not reveal the identity of the product inside (whether it is Eylea or MYL-1701P) and will be assigned in a masked fashion through the Interactive Response Technology (IRT) system. An un-masked team will identified at site, to be responsible for preparation and administration of the study drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MYL-1701P (Experimental): MYL-1701P
  Interventions: Drug: MYL-1701P
- Eylea (Active Comparator): Eylea
  Interventions: Drug: Eylea

INTERVENTIONS:
Drug: MYL-1701P — Subjects will receive intravitreal injections of MYL-1701P throughout the 52-week treatment period, with the last dose at 48 weeks.
  The additional doses may be administered in accordance with the protocol.
  Arms: MYL-1701P
Drug: Eylea — Subjects will receive intravitreal injections of Eylea throughout the 52-week treatment period, with the last dose at 48 weeks.
  The additional doses may be administered in accordance with the protocol.
  Arms: Eylea

SUMMARY:
Three hundred and twenty-four (324) eligible adult subjects with diabetes mellitus with central DME involvement to be randomized 1:1 to intravitreal treatment with MYL-1701P or Eylea®.

The primary endpoint is mean change from baseline in Best Corrected Visual Acuity (BCVA) as assessed by Early Treatment Diabetic Retinopathy Study (ETDRS) letters. Pharmacokinetics (PK) and immunogenicity to be evaluated in the subjects participating in the study.

DETAILED DESCRIPTION:
Three hundred and twenty-four (324) eligible adult subjects with diabetes mellitus with central DME involvement to be randomized 1:1 to intravitreal treatment with MYL-1701P or Eylea®. Subjects to receive the assigned treatment until Week 48.

All subjects to return to clinic every 4 weeks to assess safety, efficacy and to guide treatment. Additional visits allowed during the study as specified in the study schedule for safety and pharmacokinetic evaluation.

Pharmacokinetics (PK) and Immunogenicity to be assessed in the subjects participating in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects age ≥ 18 years.
2. Subjects have type 1 or type 2 diabetes mellitus who present with central DME involvement in the study eye.
3. The cause of decreased vision in the study eye has been attributed primarily to DME by the Investigator.
4. Subject is able to understand and voluntarily provide written informed consent to participate in the study.
5. If female of child bearing potential, the subject must have a negative serum pregnancy test at the Screening visit and a negative urine pregnancy test at baseline visit, and should not be nursing or planning a pregnancy.
6. If female, subject must be:

   1. Surgically sterilized via hysterectomy, bilateral oophorectomy, or bilateral tubal ligation; or
   2. Of childbearing potential and practicing an acceptable form of birth control (defined as the use of an intrauterine device; a barrier method, like condom, with spermicide; any form of hormonal contraceptives; or abstinence from sexual intercourse) starting 60 days prior to dosing and continuing at least 90 days following the last treatment.
   3. Of non-childbearing potential (i.e., postmenopausal for at least 1 year).
7. If male, subject must be surgically or biologically sterile. If not sterile, the subject must agree to use an acceptable form of birth control with sexual partner (as described in inclusion criteria #6b of protocol) or abstain from sexual relations during the study period and up to 90 days following the last treatment dose.
8. Subject is willing to comply with the study duration, study visits and study related procedures.

Exclusion Criteria:

1. Subjects with known hypersensitivity to aflibercept or any of the excipients
2. Subjects with current or planned use of systemic medications known to be toxic to the lens, retina or optic nerve, including deferoxamine, chloroquine/hydroxychloroquine, tamoxifen, phenothiazines and ethambutol
3. Subjects with uncontrolled hypertension defined as systolic blood pressure >160mm Hg or diastolic blood pressure > 95 mm of Hg.
4. Subjects with a history of cerebrovascular accident or myocardial infarction within 6 months of randomization.
5. Subjects with history of use of intraocular corticosteroids anytime in the past or periocular (subconjunctival, intra-scleral, sub-tenon or retrobulbar) corticosteroids within 4 months of randomization
6. Subjects who have only one functional eye, even if the eye met all other study requirements, or who have an ocular condition on the fellow eye with a poorer prognosis than the study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2021-09-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (67):
- United States (12):
  - Mylan Investigator Site, Phoenix, Arizona
  - Mylan Investigator Site, Sacramento, California
  - Mylan Investigator Site, St. Petersburg, Florida
  - Mylan Investigator Site, Winter Haven, Florida
  - Mylan Investigator Site, Augusta, Georgia
  - Mylan Investigator Site, Shawnee Mission, Kansas
  - Mylan Investigator Site, Paducah, Kentucky
  - Mylan Investigator Site, Chevy Chase, Maryland
  - Mylan Investigator Site, Ladson, South Carolina
  - Mylan Investigator Site, Nashville, Tennessee
  - Mylan Investigator Site, Abilene, Texas
  - Mylan Investigator Site, Morgantown, West Virginia
- Czechia (6):
  - Mylan Investigator Site, Prague, Vinohrady
  - Mylan Investigator Site, Hradec Králové
  - Mylan Investigator Site, Olomouc
  - Mylan Investigator Site, Pardubice
  - Mylan Investigator Site, Prague
  - Mylan Investigator Site, Zlín
- Germany (3):
  - Mylan Investigator Site, Göttingen, Lower Saxony
  - Mylan Investigator Site, Mainz, Rheinland-Pflaz
  - Mylan Investigator Site, Marburg
- Hungary (6):
  - Mylan Investigator Site, Budapest
  - Mylan Investigator Site, Debrecen
  - Mylan Investigator Site, Nyíregyháza
  - Mylan Investigator Site, Pécs
  - Mylan Investigator Site, Szeged
  - Mylan Investigator Site, Zalaegerszeg
- India (13):
  - Mylan Investigator Site, Visakhapatnam, Andhra Pradesh
  - Mylan Investigator Site, Ahmedabad, Gujarat
  - Mylan Investigator Site, Bangalore, Karnataka
  - Mylan Investigator site, Bangalore, Karnataka
  - Mylan Investigator Site, Mumbai, Maharashtra
  - Mylan Investigator Site, New Delhi, National Capital Territory of Delhi
  - Mylan Investigator Site, Bhubaneswar, Odisha
  - Mylan Investigator Site, Chandigarh, Punjab
  - Mylan Investigator Site, Jaipur, Rajasthan
  - Mylan Investigator Site, Madurai, Tamil Nadu
  - Mylan Investigator Site, Tirunelveli, Tamil Nadu
  - Mylan Investigator Site, Hyderabad, Telangana
  - Mylan Investigator Site, Noida, Uttar Pradesh
- Japan (14):
  - Mylan Investigator Site, Nagoya, Aichi-ken
  - Mylan Investigator Site, Kōriyama, Fukushima
  - Mylan Investigator Site, Sapporo, Hokkaido
  - Mylan Investigator Site, Mito, Ibaraki
  - Mylan Investigator Site, Yamato, Kanagawa
  - Mylan Investigator Site, Susono, Shizuoka
  - Mylan Investigator Site, Kofu, Yamanashi
  - Mylan Investigator Site, Fukuoka
  - Mylan Investigator Site, Fukushima
  - Mylan Investigator Site, Kagoshima
  - Mylan Investigator Site, Kumamoto
  - Mylan Investigator Site, Nagasaki
  - National Hospital Organization Osaka National Hospital, Osaka
  - Mylan Investigator Site, Saitama
- Latvia (2):
  - Mylan Investigator Site, Jelgava
  - Mylan Investigator Site, Riga
- Poland (6):
  - Mylan Investigator Site, Katowice, Silesian Voivodeship
  - Mylan Investigator Site, Tarnów, Tarnow
  - Mylan Investigator Site, Olsztyn, Warmian-Masurian Voivodeship
  - Mylan Investigator Site, Rzeszów
  - Mylan Investigator Site, Wałbrzych
  - Mylan Investigator Site, Lodz, Łódź Voivodeship
- Russia (5):
  - Mylan Investigator Site, Kazan', Tatarstan Resp.
  - Mylan Investigator Site, Moscow
  - Mylan Investigator Site, Novosibirsk
  - Mylan Investigator Site, Omsk
  - Mylan Investigator Site, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bressler SB, Barve A, Ganapathi PC, Beckmann K, Apte RS, Marcus DM, Baumane K, Agarwal S, Oleksy P, Reichstein DA, Patel SS, Ernest J, Degi R, Gupta V, Kishino G, Kamei M, Loganathan S; INSIGHT Study Group. Aflibercept Biosimilar MYL-1701P vs Reference Aflibercept in Diabetic Macular Edema: The INSIGHT Randomized Clinical Trial. JAMA Ophthalmol. 2024 Oct 1;142(10):952-960. doi: 10.1001/jamaophthalmol.2024.3458. PMID 39264599

RESULTS

PARTICIPANT FLOW:
Groups:
- MYL-1701P: MYL-1701P
  MYL-1701P: Subjects received intravitreal injections of MYL-1701P throughout the 52-week treatment period, with the last dose at 48 weeks.
  Additional doses may be administered in accordance with the protocol.
- Eylea: Eylea
  Eylea: Subjects received intravitreal injections of Eylea throughout the 52-week treatment period, with the last dose at 48 weeks.
  Additional doses may be administered in accordance with the protocol.
Period: Overall Study
Arm/Group | MYL-1701P | Eylea
Started | 179 | 176
Treated | 178 | 176
Completed | 161 | 158
Not Completed | 18 | 18

BASELINE CHARACTERISTICS:
Groups:
- MYL-1701P: MYL-1701P
  MYL-1701P: Subjects received intravitreal injections of MYL-1701P throughout the 52-week treatment period, with the last dose at 48 weeks.
  Additional doses were administered in accordance with the protocol.
- Eylea: Eylea
  Eylea: Subjects received intravitreal injections of Eylea throughout the 52-week treatment period, with the last dose at 48 weeks.
  Additional doses were administered in accordance with the protocol.
- Total: Total of all reporting groups
Arm/Group | MYL-1701P | Eylea | Total
Number analyzed (Participants) | 179 | 176 | 355
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 101 | 106 | 207
  >=65 years | 78 | 70 | 148
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.8 (8.37) | 61.6 (9.93) | 62.2 (9.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 67 | 139
  Male | 107 | 109 | 216
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 62 | 58 | 120
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 3 | 5
  White | 114 | 114 | 228
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Latvia | 9 | 9 | 18
  Hungary | 25 | 27 | 52
  United States | 32 | 31 | 63
  Czechia | 20 | 23 | 43
  Japan | 22 | 19 | 41
  Poland | 22 | 15 | 37
  Germany | 3 | 8 | 11
  India | 38 | 39 | 77
  Russia | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) at Week 8
Description: Mean change from baseline in BCVA as assessed by Early Treatment Diabetic Retinopathy Study (ETDRS) letters at week 8.
  Best Corrected Visual Acuity (BCVA) is measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the ETDRS chart, the worse the vision (or visual acuity). A positive change from baseline indicates an improvement and a negative change from baseline indicates a worsening.
Time Frame: Baseline and 8 weeks
Population: The intention-to-treat (ITT) analysis set consists of all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: BCVA letter score
Arm/Group | MYL-1701P | Eylea
Number analyzed (Participants) | 179 | 176
BCVA letter score | 6.60 (0.548) | 6.56 (0.548)
Statistical Analysis 1: Comparison: MYL-1701P vs Eylea; Test type: Equivalence — An equivalence margin of [-3, 3] letters was used to demonstrate equivalence for the difference of mean change in BCVA, from baseline to Week 8; Mean Difference (Final Values) = 0.04, 90% CI 2-sided [-1.16 to 1.24], Standard Error of Mean 0.730

2. Secondary Outcome: The Mean Change From Baseline in Central Retinal Thickness (CRT)
Description: The mean change from baseline in Central Retinal Thickness as determined by Spectral domain- Optical coherence tomography (SD-OCT) over time
Time Frame: From baseline to week 52
Population: The intention-to-treat (ITT) analysis set consists of all randomized subjects.
Measure: Mean (Standard Error); unit: Micrometer
Groups:
- MYL-1701P: MYL-1701P
  MYL-1701P: Subjects will receive intravitreal injections of MYL-1701P throughout the 52-week treatment period, with the last dose at 48 weeks.
  The additional doses may be administered in accordance with the protocol.
- Eylea: Eylea
  Eylea: Subjects will receive intravitreal injections of Eylea throughout the 52-week treatment period, with the last dose at 48 weeks.
  The additional doses may be administered in accordance with the protocol.
Arm/Group | MYL-1701P | Eylea
Number analyzed (Participants) | 179 | 176
Micrometer | -170.14 (7.198) | -167.67 (7.260)

3. Secondary Outcome: The Mean Change in BCVA
Description: Mean change from baseline in BCVA as assessed by ETDRS letters over time. Best Corrected Visual Acuity (BCVA) is measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the ETDRS chart, the worse the vision (or visual acuity). A positive change from baseline indicates an improvement and a negative change from baseline indicates a worsening
Time Frame: From baseline to week 52
Population: The intention-to-treat (ITT) analysis set consists of all randomized subjects.
Measure: Mean (Standard Error); unit: BCVA letter score
Arm/Group | MYL-1701P | Eylea
Number analyzed (Participants) | 179 | 176
BCVA letter score | 10.76 (0.619) | 10.52 (0.621)

4. Secondary Outcome: Number of Subjects Who Gained ≥15 Letters From Baseline in BCVA
Description: Number of subjects who gained ≥15 letters from baseline in BCVA, assessed in change from baseline in ETDRS letters over time
Time Frame: From baseline to week 52
Population: All randomized subjects with last observation carried forward (LOCF) value at timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | MYL-1701P | Eylea
Number analyzed (Participants) | 176 | 174
Participants | 57 | 51

5. Secondary Outcome: Number of Administrations of Study Drug Required
Description: The mean number of doses administered during the 52 weeks of study
Time Frame: From baseline to week 52
Population: The intention-to-treat (ITT) analysis set consists of all randomized subjects.
Measure: Mean (Standard Deviation); unit: Doses
Arm/Group | MYL-1701P | Eylea
Number analyzed (Participants) | 179 | 176
Doses | 8.4 (2.06) | 8.7 (1.76)

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Number of Participants with Treatment Emergent Adverse Events (Safety and tolerability)
Time Frame: From baseline to week 52
Population: Population consists of all subjects who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | MYL-1701P | Eylea
Number analyzed (Participants) | 178 | 176
Participants | 138 | 138

7. Secondary Outcome: Number of Subjects With Induced and Boosted Anti-Drug Antibodies
Description: Number of subjects with induced and boosted Anti-Drug Antibodies (ADA) (Immunogenicity)
Time Frame: From baseline to week 52
Population: All subjects who received at least one dose of study drug and have baseline and at least one post-baseline ADA results.
Measure: Count of Participants; unit: Participants
Arm/Group | MYL-1701P | Eylea
Number analyzed (Participants) | 177 | 176
Participants | 5 | 10

8. Secondary Outcome: Concentration of Aflibercept in Blood (Pharmacokinetics)
Description: Free Drug Concentration of aflibercept in blood (Pharmacokinetics)
Time Frame: 2 Days after Week 16 Injection
Population: All subjects who have signed the Informed Consent Form (ICF) for participation in Pharmacokinetics (PK) subpopulation and have at least one measured concentration of study treatment.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | MYL-1701P | Eylea
Number analyzed (Participants) | 42 | 47
ng/ml | 34.355 (30.693) | 30.758 (32.3208)

ADVERSE EVENTS:
Time Frame: Baseline to 52 Weeks
Description: Population used for analysis consist of patients treated with study drug (at least receiving one dose of MYL-1701P or Eylea)
Arm/Group | MYL-1701P | Eylea
All-Cause Mortality (participants affected / at risk) | 2/178 | 4/176
Serious Adverse Events (participants affected / at risk) | 31/178 | 23/176
Other Adverse Events (participants affected / at risk) | 53/178 | 61/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MYL-1701P (N=178) | Eylea (N=176)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 4 (4)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Atypical Pnuemonia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis Chronic (Infections and infestations) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Embolic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Thrombotic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2)
Corneal oedema (Eye disorders) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Endolymphatic hydrops (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MYL-1701P (N=178) | Eylea (N=176)
Cataract (Eye disorders) | 12 (17) | 12 (12)
Diabetic retinal oedema (Eye disorders) | 9 (9) | 10 (13)
Nasopharyngitis (Infections and infestations) | 14 (19) | 10 (10)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (3) | 9 (10)
Hypertension (Vascular disorders) | 16 (20) | 20 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT03610646/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/46/NCT03610646/SAP_001.pdf